CLINICAL TRIAL: NCT02933255
Title: Phase I/II Study of PROSTVAC in Combination With Nivolumab in Men With Prostate Cancer
Brief Title: PROSTVAC in Combination With Nivolumab in Men With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170007; 17-C-0007
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: Safety; Neoadjuvant; Prostatectomy; Immunotherapy; Vaccine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prostate-Specific Antigen; Nivolumab; Prostatectomy; Biopsy; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort (Experimental): Prostate-specific antigen (PSA)-TRICOM vaccinia (PROSTVAC)-V on week 0 followed by booster injection called PROSTVAC-F on week 2, 4, and 8. Nivolumab will be administered on week 2, 4, 6, 8 and 10. When administered on the same day, the preferred order of administration is PROSTVAC first followed by nivolumab. Participants will undergo restaging scans on week 12. If no progressive disease (PD), option to continue treatment with nivolumab every 2 weeks and PROSTVAC-F every 4 weeks until intolerance or progression. Option to extend nivolumab interval to 4 weeks for participants who remain on protocol beyond 1 year.
  Interventions: Biological: PROSTVAC-V/F; Drug: Nivolumab; Drug: Tylenol
- Neoadjuvant Cohort (Experimental): Prostate-specific antigen (PSA)-TRICOM vaccinia (PROSTVAC)-V on week 0 followed by booster injection called PROSTVAC-fowlpox (F) on 2, 4 and 8 weeks. Nivolumab will be administered on week 2, 4, and 8. When administered on the same day, the preferred order of administration is PROSTVAC first followed by nivolumab. Participants will undergo prostatectomy on week 9.
  Interventions: Biological: PROSTVAC-V/F; Drug: Nivolumab; Procedure: Prostatectomy; Procedure: Biopsy; Drug: Tylenol

INTERVENTIONS:
Biological: PROSTVAC-V/F — PROSTVAC-V (vaccinia) will be administered subcutaneously in an extremity (e.g., thigh) at a dose of 2x10^8 infectious units. PROSTVAC-F (fowlpox) will be administered subcutaneously in an extremity (e.g., thigh) at a dose of 1x10^9 infectious units.
  Other Names: Prostate-specific antigen (PSA)-TRICOM vaccinia fowlpox (PROSTVAC-V/F)
Drug: Nivolumab — Nivolumab is to be administered as a flat dose over approximately 30-minutes via intravenous (IV) infusion.
  Other Names: Opdivo
Procedure: Prostatectomy — Participants in the neoadjuvant cohort will undergo a radical prostatectomy in week 9. (If surgery is scheduled earlier than 9 weeks after initial dosing, the 6 and 8 week dosing may be skipped, and surgery may be done as early as week 5.)
  Arms: Neoadjuvant Cohort
Procedure: Biopsy — A baseline biopsy is performed for participants in the neoadjuvant cohort that do not have a previous collection of biopsy material.
  Arms: Neoadjuvant Cohort
Drug: Tylenol — Participants who experience aches or fever after vaccination may take Tylenol as directed.
  Other Names: Acetaminophen

SUMMARY:
Background:

The immune system is the cells and organs in the body that recognize and fight infection and cancer. The prostate specific antigen (PSA)/TRICOM (PROSTVAC) vaccine might teach the immune system to find and kill certain prostate cancer cells. Nivolumab is a drug that allows the immune system to fight tumors. It might help PROSTVAC work better.

Objective:

To test the safety and effectiveness of the combination of PROSTVAC and nivolumab. To test this for people with castration resistant prostate cancer and then for other people with localized prostate cancer who are candidates for surgical removal of the prostate.

Eligibility:

Men ages 18 and older with prostate cancer

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Electrocardiogram

Bone scan

Computed tomography (CT) scan or magnetic resonance imaging (MRI)

Tumor sample. This may be from a previous procedure.

All participants will get a combination of the study drugs over 8 weeks. They will have 1 visit for the initial injection then 3 booster injection / nivolumab infusion visits. Blood will be tested at these visits.

Over the next 4 weeks, some participants will have:

An exam of the large intestine through the rectum.

CT and bone scans

Standard hormonal treatment

Option to continue treatment every 3 weeks if their disease does not get worse. They will have scans every 12 weeks.

Other participants will have surgery to remove the prostate in week 9.

Participants will have a safety visit about a month after their last treatment. This will include a physical exam, blood tests, and possibly scans.

If their cancer progresses, participants will leave the study and may enroll in a long-term follow-up study. They will be contacted once a year to ask about their cancer and treatment.

DETAILED DESCRIPTION:
Background:

Immune checkpoint inhibitors interfere with the immune systems autoregulatory mechanisms, allowing for a potentially expanded and prolonged T-cell response with the possibility of greater antitumor effects.

Nivolumab is a fully human Immunoglobulin G4 (IgG4) monoclonal antibody that targets the programmed cell death protein 1 (PD-1) protein. Specifically, the antibody binds to the PD-1 receptor and blocks its interaction with programmed death-ligand 1 (PD-L1) and programmed cell death 1 ligand 2 (PD-L2), thereby releasing PD-1 pathway-mediated inhibition of the immune response, including anti-tumor immune response.

PROSTVAC (developed by the National Cancer Institute [NCI] and licensed to Bavarian Nordic Immunotherapeutics, Mountain View, California (CA) is a therapeutic cancer vaccine for prostate cancer. Early studies have demonstrated immunologic efficacy and suggested clinical benefit. A phase III trial has completed accrual.

A previous study combining the immune checkpoint inhibitor ipilimumab and PROSTVAC suggested greater efficacy than PROSTVAC alone. Additional studies have demonstrated the potential efficacy of immunologic combination therapy with the immune checkpoint inhibitor nivolumab.

This study will aim to evaluate the impact of the combination of PROSTVAC and the immune checkpoint inhibitor nivolumab on the tumor microenvironment focusing on immune cell infiltration as the primary endpoint.

United States (US)-MRI imaging technology will be employed to sample the tumor before treatment and after radical prostatectomy.

The findings from this study could serve as the basis for future studies with this combination in this population of participants and more advanced disease.

Objectives:

Safety (For castration resistant prostate cancer (CRPC) lead-in cohort)

Evaluate changes in T-cell infiltration in the tumor after neoadjuvant treatment with PROSTVAC and nivolumab, relative to changes seen in a phase 2 trial with PROSTVAC alone in the neoadjuvant setting- NCT02153918 (For the neoadjuvant cohort).

Eligibility:

Participants must have histopathological documentation of adenocarcinoma of the prostate prior to starting this study and evaluable biopsy tissue (e.g., unstained slides or blocks) available for analysis.

For the castration resistant lead in cohort, if histopathological documentation is unavailable, a rising prostate specific antigen (PSA) and a clinical course consistent with prostate cancer would be acceptable.

Participants must have a performance status of 0 to 1 according to the Eastern Cooperative Oncology Group (ECOG) criteria.

Hematological eligibility parameters (within 16 days of starting therapy):

Granulocyte count 1,500/mm^3

Platelet count 100,000/mm^3

Hemoglobin (Hgb) >= 8 g/dL

Biochemical eligibility parameters (within 16 days of starting therapy):

Hepatic function: Bilirubin < 1.5 mg/dl (OR in participants with Gilbert's syndrome, total bilirubin <= 3.0 mg/dL), aspartate aminotransferase (AST) and alanine transaminase (ALT) <= 2.5 times upper limit of normal.

Creatinine <= 1.5 X ULN

Design:

The primary focus of this study will be to evaluate PROSTVAC and nivolumab in the neoadjuvant setting.

Lead-in cohort evaluating the safety and tolerability of this combination in the castration resistant setting (CRPC cohort)

Following this lead-in cohort in the CRPC setting, we will enroll a cohort in the neoadjuvant setting evaluating the combination of PROSTVAC and nivolumab.

The lead-in safety cohort will require 10 participants and the neoadjuvant cohort will require 17 evaluable participants. In order to allow for a small number of inevaluable participants, the accrual ceiling will be set to 29 participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

For the neoadjuvant cohort, patients must have histopathological documentation of adenocarcinoma of the prostate prior to starting this study and evaluable biopsy tissue (e.g., unstained slides or blocks) available for analysis. If evaluable tissue is not available, the patient must agree to undergo a pre-vaccination prostate biopsy on study. For the castration-resistant prostate cancer (CRPC) lead in cohort, if histopathological documentation is unavailable, a rising prostate specific antigen (PSA) and a clinical course consistent with prostate cancer would be acceptable.

* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of PROSTVAC in combination with nivolumab, ipilimumab or both in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants must not have other active invasive malignancies within the past 2 years (with the exception, of non-melanoma skin cancers) (for CRPC cohort only).
* Participants must be willing to travel to the study site for follow-up visits
* All participants who have received prior vaccination with vaccinia virus (for smallpox immunization) must not have a history of serious adverse reaction to the vaccine.
* The effects of PROSTVAC in combination nivolumab, ipilimumab or both on the developing human fetus are unknown. For this reason, men must agree to use adequate contraception (abstinence, vasectomy) or female partner must use (intrauterine device (IUD), hormonal [birth control, pills, injections, or implants], tubal ligation] prior to study entry and for up to 7 months after the last dose.
* Participants must understand and sign informed consent that explains the neoplastic nature of their disease, the procedures to be followed, the experimental nature of the treatment, alternative treatments, potential risks and toxicities, and the voluntary nature of participation.
* Participants must have normal organ and marrow function as defined below:

  * hemoglobin greater than or equal to 8 g/dL
  * granulocytes greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin < 1.5 mg/dL (or less than or equal to 3.0 mg/dL in patients with Gilbert syndrome)
  * Aspartate aminotransferase (AST)serum glutamic oxaloacetic transaminase (SGOT)(SGOT)/alanine transaminase (ALT)serum glutamic-pyruvic transaminase (SGPT) less than or equal to 2.5 X institutional upper limit of normal
  * creatinine less than or equal to 1.5 X ULN
* For the lead in cohort:

  * Castrate testosterone level (<50ng/dl or 1.7nmol /L)
  * Progressive disease at study entry defined as one or more of the following criteria occurring in the setting of castrate levels of testosterone:

    * Radiographic progression defined as any new or enlarging bone lesions or growing lymph node disease, consistent with prostate cancer OR
    * PSA progression defined by sequence of rising values separated by >1 week (2 separate increasing values over a minimum of 2ng/ml (Prostate Cancer Clinical Trials Working Group (PCWG2) PSA eligibility criteria). If participants had been on flutamide, PSA progression is documented 4 weeks or more after withdrawal. For patients on bicalutamide or nilutamide disease progression is documented 6 or more weeks after withdrawal.
  * Participants must agree to continuation of androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone agonist/antagonist or bilateral orchiectomy
* For all neoadjuvant cohorts:

  * Participants must be a surgical candidate for radical prostatectomy based on standard workup of PSA, biopsy results, and if necessary supplemental imaging.
  * Participants must have chosen radical prostatectomy as their definitive treatment of choice for management of their prostate cancer.
  * No systemic steroid or steroid eye drop use within 2 weeks prior to initiation of experimental therapy. Limited doses of systemic steroids to prevent intravenous (IV) contrast, allergic reaction or anaphylaxis (in patients who have known contrast allergies) are allowed.

EXCLUSION CRITERIA:

* Prior splenectomy.
* The recombinant vaccinia vaccine should not be administered if the following apply to either recipients or, for at least 3 weeks after vaccination, their close household contacts (Close household contacts are those who share housing or have close physical contact):

  * persons with active or a history of eczema or other eczematoid skin disorders
  * those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne or other open rashes or wounds) until condition resolves
  * pregnant or nursing women; children under 3 years of age
* Participants should have no evidence, as listed below, of being immunocompromised:

  * Human immunodeficiency virus (HIV) positivity due to the potential for decreased tolerance and risk for severe side effects.
  * Hepatitis B or C positivity.
* Concurrent use of systemic steroids or steroid eye drops. This is to avoid immunosuppression which may lead to potential complications with vaccinia (priming vaccination). Nasal, topical, or inhaled steroid use is permitted.
* Participants with known allergy to eggs or to compounds with a similar chemical or biologic composition to PROSTVAC, ipilimumab or nivolumab.
* No prior immune checkpoint inhibitors (e.g., anti-cytotoxic T-lymphocyte associated protein 4 (CTLA4), anti-programmed cell death protein 1 (PD-1) or anti-programmed death-ligand 1 (PDL1) are allowed.
* Other serious intercurrent illness.
* Participants with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment) or New York Heart Association class II-IV congestive heart failure.
* Participants with significant autoimmune disease that is active or potentially life threatening if activated.
* Participants with clinically significant cardiomyopathy requiring treatment.
* Participants with ongoing toxicities related to prior therapies targeting T cell coregulatory proteins (immune checkpoints) such as anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody are excluded
* No transfusion of blood or blood products within 2 weeks and no granulocyte colony stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 2 weeks prior to initiations of experimental therapy.
* Contraindication to biopsy or prostatectomy (for sequential neoadjuvant cohorts only):

  * Bleeding disorders
  * Artificial heart valve
  * Prothrombin time (PT)/partial thromboplastin time (PTT) greater than or equal to 1.5 in participants not taking anticoagulation. Participants on anticoagulation (e.g., enoxaparin, oral anticoagulants) are eligible regardless of PT/PTT. Prior to biopsy, anticoagulation will be held per standard practice.
* For participants with localized prostate cancer contraindication to magnetic resonance imaging (MRI):

  * Participants weighing >136 kilograms (weight limit for the scanner tables)
  * Allergy to magnetic resonance (MR) contrast agent
  * Participants with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices
* History of radiation proctitis (for lead-in CRPC cohort only)

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Lassoued W, Madan RA, Xue E, Burnett D, Canubas KD, Bailey S, Marte JL, Tsai YT, Donahue RN, Turkbey IB, Papanicolau-Sengo A, Williams M, Hankin A, Manukyan M, Manu M, Kang Z, Pritchard C, Dahut W, Karzai F, Schlom J, Sater S, Pinto P, Gulley JL. Programmed death-1 inhibition increases vaccine-induced T-cell infiltration in patients with prostate cancer. J Immunother Cancer. 2025 Jun 22;13(6):e010851. doi: 10.1136/jitc-2024-010851. PMID 40550568
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0007.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort | Neoadjuvant Cohort
Started | 12 | 12
Follow Up Period Completed | 11 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Discontinued due to study closure. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort | Neoadjuvant Cohort | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 9 | 12
  >=65 years | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.48 (7.42) | 60.93 (6.53) | 66.2 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Important Immune-related Adverse Events (for the Lead-In Cohort)
Description: Clinically important immune-related adverse events were defined as grade 3 or above inflammation requiring steroids or anti cytokine therapy or not resolving to grade 1 or less within 28 days. These immune-related adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 3 is severe, grade 4 is life-threatening, and grade 5 is death related to adverse event.
Time Frame: From treatment start throughout study completion, an average of 1.4 years.
Population: *2 out of 7 immune related adverse events (irAEs) occurred during administration of both ipilimumab and nivolumab, before a protocol amendment was performed and eliminated ipilimumab from the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort
Number analyzed (Participants) | 12
Participants
  Grade 3 irAE colitis | 1
  Grade 3 irAE hemorrhagic cystitis | 1
  Grade 3 irAE hepatitis (alanine aminotransferase (ALT) increase) | 1
  Grade 3 irAE maculopapular rash | 1
  Grade 3 irAE mucositis oral | 1
  Grade 4 autoimmune diabetes (hyperglycemia) | 1
  Grade 4 irAE myositis (CPK increase) | 1
  Grade 4 irAE hepatitis (alanine aminotransferase (ALT)/aspartate aminotransferase (AST) increase) | 1
  Grade 5 irAE | 0

2. Primary Outcome: Changes in T-cell Infiltration in the Tumor After Neoadjuvant Treatment (Only for the Neoadjuvant Cohort)
Description: Changes in T-cell infiltration in the tumor after neoadjuvant treatment with PROSTVAC and nivolumab, is defined as difference in density of cytotoxic T lymphocytes (CD8 T) cells and clusters of differentiation 4 (CD4 T) cells infiltrate from baseline to post-treatment (radical prostatectomy performed at week 9), calculated utilizing computer automated staining analysis. The analysis was done per tissue compartment (normal region, intra-tumoral and invasive margin). We hypothesized an increase in T cell infiltration after treatment. Statistically significant changes in T-cell infiltration are those with p<0.05; to 0.05. The changes are not statistically significant.
Time Frame: From baseline to radical prostatectomy (approximately week 9)
Measure: Median (Inter-Quartile Range); unit: Cell/mm^2 of tissue
Arm/Group | Neoadjuvant Cohort
Number analyzed (Participants) | 12
Cell/mm^2 of tissue
  CD8+ T cell in the total tissue at baseline | 64.02 [41.2 to 133.7]
  CD8+ T cell in the total tissue at prostatectomy at week 9 | 154.3 [80.2 to 312.3]
  CD8+ T cell in the center of the tumor at baseline | 57.9 [26.5 to 103.8]
  CD8+ T cell in the center of the tumor at prostatectomy at week 9 | 110.5 [58.3 to 221]
  CD8+ T cell in the invasive margin at baseline | 56.4 [49.3 to 88.5]
  CD8+ T cell in the invasive margin at prostatectomy at week 9 | 304 [136.5 to 522.5]
  CD8+ T cell in the normal region at baseline | 99.15 [58.2 to 207.8]
  CD8+ T cell in the normal region at prostatectomy at week 9 | 124.5 [80.5 to 231.5]
  CD4+ T cell helper in the total tissue at baseline | 114.4 [61.1 to 184.9]
  CD4+ T cell helper in the total tissue at prostatectomy at week 9 | 478.8 [319.3 to 632.1]
  CD4+ T cell helper in the center of the tumor at baseline | 109.5 [70.5 to 149.7]
  CD4+ T cell in the center of the tumor at prostatectomy at week 9 | 394.5 [114.3 to 676]
  CD4+ T cell helper in the invasive margin at baseline | 161 [59.8 to 206.4]
  CD4+ T cell helper in the invasive margin at prostatectomy at 9 weeks | 672.5 [587 to 1225.3]
  CD4+ T cell helper in the normal region at baseline | 57.4 [37.5 to 113.4]
  CD4+ T cell helper in the normal region at prostatectomy at week 9 | 246.5 [97 to 361.3]
Statistical Analysis 1: Comparison: Neoadjuvant Cohort; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+T cell infiltration within the total tissue at time of prostatectomy compared to baseline
Statistical Analysis 2: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.04, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+T cell infiltration in the center of the tumor at time of prostatectomy compared to baseline
Statistical Analysis 3: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.002, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+T cell infiltration in the invasive margin at time of prostatectomy compared to baseline
Statistical Analysis 4: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.46, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+T cell infiltration in the normal region at time of prostatectomy compared to baseline
Statistical Analysis 5: Comparison: Neoadjuvant Cohort; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4 T cell helper infiltration in the total tissue at time of prostatectomy compared to baseline
Statistical Analysis 6: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.016, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4 T cell helper infiltration in the center of the tumor at time of prostatectomy compared to baseline
Statistical Analysis 7: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.002, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4 T cell helper infiltration in the invasive margin at time of prostatectomy compared to baseline
Statistical Analysis 8: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.38, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4 T cell helper infiltration in the normal region at time of prostatectomy compared to baseline

3. Secondary Outcome: Number of Participants With Clinically Important Immune-related Adverse Events (Only for Neoadjuvant Cohort)
Description: Clinically important immune-related adverse events were defined as grade 3 or above inflammation requiring steroids or anti cytokine therapy or not resolving to grade 1 or less within 28 days. These immune-related adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 3 is severe, grade 4 is life-threatening, and grade 5 is death related to adverse events.
Time Frame: From baseline throughout study completion, an average of 20 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Cohort
Number analyzed (Participants) | 12
Participants | 0

4. Secondary Outcome: Changes in Soluble Immune Mediating Factors (Soluble Cluster of Differentiation 27 (sCD27) in Sera
Description: Changes in soluble immune mediating factors were defined as differences in sCD27 concentration between pre- and post-treatment samples and were measured by enzyme-linked immunosorbent assay (ELISA) and Mesoscale Assay. P values were calculated using the Wilcoxon Signed Rank Test. We hypothesized an increase in sCD27 after treatment. Statistically significant changes in soluble analyzes are those with p<0.05; to 0.05 means no statistically significant changes.
Time Frame: Week 4, week 10, and week 20 after therapy compared to baseline
Measure: Median (Inter-Quartile Range); unit: U/mL
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort | Neoadjuvant Cohort
Number analyzed (Participants) | 12 | 12
U/mL
  sCD27 at baseline | 98.6 [85.6 to 122.5] | 77.2 [59.8 to 98.9]
  sCD27 week 4 | 127.9 [85 to 164] | 80.2 [71.4 to 109.5]
  sCD27 week 10 | 108.8 [90.2 to 138.3] | 82 [70.1 to 102.8]
  SCD27 week 20 | 131.9 [95.5 to 141.2] | 81 [68.3 to 95.5]
Statistical Analysis 1: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other — The reported p-value is representative of changes in soluble factors at 4 weeks of therapy compared to baseline in the lead-in metastatic castration-resistant prostate cancer (mCRPC) cohort; p = 0.064, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Neoadjuvant Cohort; Test type: Other — The reported p-value is representative of changes in soluble factors at 4 weeks of therapy compared to baseline in the neoadjuvant cohort; p = 0.001, Wilcoxon Signed Rank Test
Statistical Analysis 3: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.003, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in soluble factors at 10 weeks of therapy compared to baseline in the lead-in metastatic castration-resistant prostate cancer (mCRPC) cohort
Statistical Analysis 4: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.003, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in soluble factors at 10 weeks of therapy compared to baseline in the neoadjuvant cohort
Statistical Analysis 5: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.004, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in soluble factors at 20 weeks of therapy compared to baseline in the lead-in metastatic castration-resistant prostate cancer (mCRPC) cohort
Statistical Analysis 6: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.004, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in soluble factors at 20 weeks of therapy compared to baseline in the neoadjuvant cohort

5. Secondary Outcome: Changes in Soluble Immune Mediating Factors (Tumor Necrosis Factor Alpha (TNFα) and Interleukin 10 (IL-10) in Sera
Description: Changes in soluble immune mediating factors were defined as differences in TNFα, and IL-10 concentration between pre- and post-treatment samples and were measured by enzyme-linked immunosorbent assay (ELISA) and Mesoscale Assay. P values were calculated using the Wilcoxon Signed Rank Test. We hypothesized an increase in TNFα and IL-10 after treatment. Statistically significant changes in soluble analyzes are those with p<0.05, p0.05 means the changes are not statistically significant.
Time Frame: Week 4, week 10, and week 20 after therapy compared to baseline
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort | Neoadjuvant Cohort
Number analyzed (Participants) | 12 | 12
pg/mL
  TNFα Baseline | 2.8 [2.5 to 3.9] | 2.5 [1.6 to 3]
  TNFα Week 4 | 3.5 [3.1 to 4.9] | 2.7 [2.3 to 4.1]
  TNFα Week 10 | 3 [2.7 to 4.9] | 2.8 [2.4 to 3.2]
  TNFα Week 20 | 3.4 [3 to 4.1] | 2.4 [2.1 to 3.1]
  IL-10 Baseline | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.3]
  IL-10 Week 4 | 0.6 [0.4 to 0.8] | 0.5 [0.3 to 0.6]
  IL-10 Week 10 | 0.5 [0.3 to 1] | 0.4 [0.3 to 0.6]
  IL-10 Week 20 | 0.5 [0.4 to 0.9] | 0.5 [0.3 to 0.6]
Statistical Analysis 1: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.002, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in TNFα at 4 weeks of therapy compared to baseline in the lead-in metastatic castration-resistant prostate cancer (mCRPC) cohort
Statistical Analysis 2: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.042, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in TNFα at 4 weeks of therapy compared to baseline in the neoadjuvant cohort
Statistical Analysis 3: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.233, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in TNFα at 10 weeks of therapy compared to baseline in the lead-in metastatic castration-resistant prostate cancer (mCRPC) cohort
Statistical Analysis 4: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.052, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in TNFα at 10 weeks of therapy compared to baseline in the neoadjuvant cohort
Statistical Analysis 5: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.055, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in TNFα at 20 weeks of therapy compared to baseline in the lead-in metastatic castration-resistant prostate cancer (mCRPC) cohort
Statistical Analysis 6: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.203, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in TNFα at 20 weeks of therapy compared to baseline in the neoadjuvant cohort
Statistical Analysis 7: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p < 0.001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in IL-10 at 4 weeks of therapy compared to baseline in the lead-in metastatic castration-resistant prostate cancer (mCRPC) cohort
Statistical Analysis 8: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.034, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in IL-10 at 4 weeks of therapy compared to baseline in the neoadjuvant cohort
Statistical Analysis 9: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p < 0.001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in IL-10 at 10 weeks of therapy compared to baseline in the lead-in metastatic castration-resistant prostate cancer (mCRPC) cohort
Statistical Analysis 10: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.034, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in IL-10 at 10 weeks of therapy compared to baseline in the neoadjuvant cohort
Statistical Analysis 11: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.004, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in IL-10 at 20 weeks of therapy compared to baseline in the lead-in metastatic castration-resistant prostate cancer (mCRPC) cohort
Statistical Analysis 12: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.129, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in IL-10 at 20 weeks of therapy compared to baseline in the neoadjuvant cohort

6. Secondary Outcome: Percent Change of Tumor Cells Expressing Programmed Death-ligand 1 (PDL-1) (for the Neo-adjuvant Cohort)
Description: Changes in PD-L1 expression is defined as changes in density of cells positive for PDL1 and was analyzed by immunohistochemistry staining using the clone 22C3. Placenta tissue was used as a positive control. Previous studies have shown that high PDL1 expression is associated with poor clinical outcomes in prostate cancer participants. An increase of PDL1 after immunotherapy could indicate a resistance of the tumor to the treatment. Values can go from 0 to 100. 50% of Tumor cells is considered positive for PDL1. The sample will be considered positive if at least 1% or tumor cells express PDL1.
Time Frame: Baseline (biopsy before first PROSTVAC administration) and at time of radical prostatectomy (on week 9)
Measure: Mean (Standard Deviation); unit: Percent change in cell/mm^2 of tissue
Arm/Group | Neoadjuvant Cohort
Number analyzed (Participants) | 12
Percent change in cell/mm^2 of tissue
  Baseline | 0 (0)
  Time of prostatectomy (week 9) | 0.07 (0.16)

7. Secondary Outcome: Changes in Immune Cell Subsets in the Peripheral Blood
Description: Peripheral blood samples were collected at baseline and after treatment start via apheresis and cryopreserved peripheral blood mononucleate cells (PBMCs) were analyzed through multicolor flow cytometry to assess cell subsets, i.e. cluster of differentiation 4 (CD4+) T cells, cytotoxic T cells (CD8+) T cells, Tregs, B cells, Natural Killer (NK) cells, NK-T cells, conventional Dendritic Cells (cDCs), plasmocytoid DCs (pDCs), myeloid-derived suppressor cells (MDSCs), and monocytes and refined subsets related to their maturation/function. P values were calculated using the Wilcoxon Signed Rank Test. Statistically significant changes in immune cell subsets are defined as those with p<0.05 and >50% of participants having a >25% change in a given subset.
Time Frame: Week 4 and week 10 after therapy compared to baseline.
Measure: Median (Inter-Quartile Range); unit: percentage of PBMC's
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort | Neoadjuvant Cohort
Number analyzed (Participants) | 12 | 12
percentage of PBMC's
  CD4+ T cells Baseline | 33.4 [24.5 to 42.9] | 27 [21.9 to 35.7]
  CD4+ T cells week 4 post treatment | 27.2 [24 to 41.5] | 20.3 [16.4 to 29]
  CD4+ T cells week 10 post treatment | 24.5 [20.5 to 38] | 25.4 [23.6 to 36.1]
  CD8+ T cells Baseline | 11.7 [8.4 to 22.1] | 10.4 [9.2 to 14.1]
  CD8+ T cells week 4 post treatment | 11 [9.5 to 19] | 9.4 [7 to 16]
  CD8+ T cells week 10 post treatment | 10.6 [7.9 to 20.4] | 10.8 [9.8 to 12.6]
  Treg cells Baseline | 0.9 [0.6 to 1] | 0.9 [0.8 to 1.1]
  Treg cells week 4 post treatment | 1.1 [0.9 to 1.4] | 1 [0.7 to 1.1]
  Treg cells week 10 post treatment | 0.6 [0.4 to 1.1] | 0.9 [0.7 to 1.3]
  cDC cells Baseline | 0.2 [0.1 to 0.4] | 0.5 [0.3 to 0.6]
  cDC cells week 4 post treatment | 0.2 [0.1 to 0.3] | 0.4 [0.3 to 0.6]
  cDC cells week 10 post treatment | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.5]
  Monocytes Baseline | 6.8 [3 to 13.4] | 12.5 [7.7 to 18]
  Monocytes week 4 post treatment | 7.5 [3.7 to 11.3] | 14.6 [9.6 to 22.4]
  Monocytes week 10 post treatment | 6.2 [3.8 to 15.9] | 10.9 [6.1 to 15.2]
  CD4+ki67+ T cells Baseline | 0.9 [0.7 to 1] | 0.5 [0.4 to 0.7]
  CD4+ki67+ T cells week 4 post treatment | 1.3 [1 to 1.9] | 0.6 [0.5 to 1]
  CD4+ki67+ T cells week 10 post treatment | 0.9 [0.7 to 1.2] | 0.6 [0.5 to 0.8]
  CD4+EM ki67+ T cells Baseline | 0.6 [0.4 to 0.7] | 0.4 [0.3 to 0.5]
  CD4+EM ki67+ T cells week 4 post treatment | 0.8 [0.7 to 1.3] | 0.5 [0.4 to 0.8]
  CD4+EM ki67+ T cells week 10 post treatment | 0.7 [0.5 to 0.9] | 0.5 [0.4 to 0.6]
  CD4+ ICOS+ T cells Baseline | 2.6 [2 to 4] | 2 [1.6 to 2.5]
  CD4+ ICOS+ T cells week 4 post treatment | 3.8 [2.8 to 5.3] | 2.3 [1.8 to 3.8]
  CD4+ ICOS+ T cells week 10 post treatment | 2.2 [1.7 to 2.9] | 2.3 [1.9 to 3.1]
  CD8+ ki67+ T cells Baseline | 0.2 [0.2 to 0.3] | 0.2 [0.1 to 0.3]
  CD8+ ki67+ T cells week 4 post treatment | 0.5 [0.3 to 0.9] | 0.2 [0.2 to 0.5]
  CD8+ ki67+ T cells week 10 post treatment | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.3]
  Treg ICOS+ cells Baseline | 0.5 [0.4 to 0.6] | 0.4 [0.3 to 0.5]
  Treg ICOS+ cells week 4 post treatment | 0.7 [0.5 to 0.9] | 0.5 [0.3 to 0.6]
  Treg ICOS+ cells week 10 post treatment | 0.4 [0.2 to 0.6] | 0.5 [0.3 to 0.6]
  NK ki67+ cells Baseline | 0.7 [0.5 to 0.8] | 0.5 [0.3 to 0.8]
  NK ki67+ cells week 4 post treatment | 1 [0.6 to 1.7] | 0.5 [0.3 to 0.8]
  NK ki67+ cells week 10 post treatment | 0.8 [0.4 to 1.1] | 0.4 [0.3 to 0.7]
  NK NKG2D+ cells Baseline | 1 [0.5 to 1.3] | 1.2 [1 to 2.2]
  NK NKG2D+ cells week 4 post treatment | 1.7 [1 to 2] | 1.6 [0.8 to 3.1]
  NK NKG2D+ cells week 10 post treatment | 1.2 [0.6 to 1.8] | 2.3 [1 to 3.2]
  NK NKp46+ cells Baseline | 2.5 [2.1 to 3] | 2 [1.2 to 2.5]
  NK NKp46+ cells week 4 post treatment | 3.3 [2.6 to 4.3] | 2.4 [1.5 to 2.7]
  NK NKp46+ cells week 10 post treatment | 3.1 [2.2 to 3.5] | 1.8 [1.1 to 2.7]
  CD8+ naive T cells Baseline | 3.3 [0.7 to 4.8] | 2.2 [1.5 to 2.8]
  CD8+ naive T cells week 4 post treatment | 2.6 [0.7 to 4.7] | 1.7 [1 to 2.4]
  CD8+ naive T cells week 10 post treatment | 2.3 [0.7 to 4.6] | 2.1 [1.6 to 2.5]
  CD8+ CM T cells Baseline | 0.3 [0.2 to 0.4] | 0.4 [0.2 to 0.6]
  CD8+ CM T cells week 4 post treatment | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.5]
  CD8+ CM T cells week 10 post treatment | 0.2 [0.1 to 0.3] | 0.4 [0.3 to 0.5]
  gMDSC Baseline | 0 [0 to 0.1] | 0 [0 to 0.1]
  gMDSC week 4 post treatment | 0 [0 to 0.1] | 0.2 [0 to 0.2]
  gMDSC week 10 post treatment | 0 [0 to 0.1] | 0.1 [0 to 0.2]
  Intermediate monocytes Baseline | 0.2 [0.1 to 0.7] | 0.4 [0.3 to 0.7]
  Intermediate monocytes week 4 post treatment | 0.4 [0.1 to 0.8] | 0.7 [0.5 to 1.8]
  Intermediate monocytes week 10 post treatment | 0.2 [0.2 to 0.6] | 0.5 [0.3 to 0.7]
  Non-classical monocytes Baseline | 0.7 [0.2 to 1.3] | 0.8 [0.5 to 1.2]
  Non-classical monocytes week 4 post treatment | 0.9 [0.2 to 1.6] | 1.6 [0.9 to 3]
  Non-classical monocytes week 10 post treatment | 0.4 [0.3 to 1.2] | 0.9 [0.6 to 1.5]
  CD4+ CM T cells Baseline | 10 [7.3 to 13.6] | 9.3 [6.7 to 11.2]
  CD4+ CM T cells week 4 post treatment | 7.5 [4.7 to 10.8] | 5.9 [4.4 to 8.6]
  CD4+ CM T cells week 10 post treatment | 7.6 [3.3 to 9.5] | 9 [7.1 to 9.9]
  CD4+ naive T cells Baseline | 9 [3.6 to 13.9] | 6.7 [4.7 to 9.8]
  CD4+ naive T cells week 4 post treatment | 8.5 [3.9 to 16.6] | 4.7 [3.5 to 7.4]
  CD4+ naive T cells week 10 post treatment | 8.8 [3.3 to 14.8] | 5.7 [3.9 to 12.8]
Statistical Analysis 1: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.339, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ T cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 2: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.037, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ T cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 3: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.009, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ T cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 4: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.844, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ T cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 5: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.204, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ T cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 6: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.084, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ T cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 7: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.042, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ T cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 8: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.688, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ T cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 9: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p < 0.001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in Treg cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 10: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.733, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in Treg cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 11: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.519, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in Treg cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 12: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.695, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in Treg cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 13: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.034, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in cDC cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 14: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.301, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in cDC cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 15: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.38, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in cDC cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 16: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.014, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in cDC cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 17: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.791, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in monocytes at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 18: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.042, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in monocytes at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 19: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.424, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in monocytes at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 20: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.77, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in monocytes at week 10 post treatment compared to baseline in the lead-in neoadjuvant cohort
Statistical Analysis 21: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ki67+ T cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 22: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.105, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ki67+ T cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 23: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.622, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ki67+ T cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 24: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.313, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ki67+ T cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 25: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p < 0.001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ EM ki67+ T cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 26: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.049, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ EM ki67+ T cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 27: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.47, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ EM ki67+ T cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 28: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.313, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ EM ki67+ T cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 29: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ ICOS+ T cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 30: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.092, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ ICOS+ T cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 31: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.176, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ ICOS+ T cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 32: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.232, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ ICOS+ T cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 33: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p < 0.001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ ki67+ T cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 34: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.131, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ ki67+ T cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 35: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.424, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ ki67+ T cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 36: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.438, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ ki67+ T cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 37: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p < 0.001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in Treg ICOS+ cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 38: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.151, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in Treg ICOS+ cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 39: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.569, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in Treg ICOS+ cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 40: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.105, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in Treg ICOS+ cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 41: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.012, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK ki67+ cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 42: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.677, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK ki67+ cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 43: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.424, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK ki67+ cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 44: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.432, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK ki67+ cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 45: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.016, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK NKG2D+ cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 46: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.733, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK NKG2D+ cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 47: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.519, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK NKG2D+ cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 48: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.557, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK NKG2D+ cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 49: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.034, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK NKp46+ cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 50: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.092, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK NKp46+ cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 51: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.733, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK NKp46+ cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 52: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.922, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in NK NKp46+ cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 53: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.176, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ naive T cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 54: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.049, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ naive T cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 55: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.001, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ naive T cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 56: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.563, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ naive T cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 57: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.012, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ CM T cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 58: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.084, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ CM T cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 59: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.016, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ CM T cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 60: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.688, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD8+ CM T cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 61: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.38, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in gMDSC at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 62: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.021, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in gMDSC at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 63: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.91, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in gMDSC at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 64: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.084, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in gMDSC at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 65: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.151, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in intermediate monocytes at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 66: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.042, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in intermediate monocytes at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 67: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.424, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in intermediate monocytes at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 68: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.846, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in intermediate monocytes at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 69: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.339, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in non-classical monocytes at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 70: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.012, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in non-classical monocytes at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 71: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.622, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in non-classical monocytes at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 72: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.492, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in non-classical monocytes at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 73: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.11, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ CM T cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 74: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.02, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ CM T cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 75: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.052, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ CM T cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 76: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.844, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ CM T cells at week 10 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 77: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p > 0.999, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ naive T cells at week 4 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 78: Comparison: Neoadjuvant Cohort; Test type: Other; p = 0.049, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ naive T cells at week 4 post treatment compared to baseline in the neoadjuvant cohort
Statistical Analysis 79: Comparison: Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort; Test type: Other; p = 0.339, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ naive T cells at week 10 post treatment compared to baseline in the lead-in metastatic castration-resistant prostate cancer cohort
Statistical Analysis 80: Comparison: Neoadjuvant Cohort; Test type: Other; p > 0.999, Wilcoxon Signed Rank Test — The reported p-value is representative of changes in CD4+ naive T cells at week 10 post treatment compared to baseline in the neoadjuvant cohort

8. Secondary Outcome: Changes in Circulating Tumor Cells (CTCs) Levels
Description: Blood samples will be collected at baseline and after treatment, and aliquoted onto slides and examined, cytokeratin-positive/lymphocyte common antigen (CD45)-negative cells with an intact nucleus and a malignancy-consistent morphology will be identified as CTCs, and their exact positions on the slides recorded.
Time Frame: At baseline and at week 9
Population: This analysis was not performed because the technology developed by Epic Sciences was still in development, thus samples were not sent to the off-site center to perform analysis.
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With a Pathologic Complete Response (pCR) (Only for Neoadjuvant Cohort)
Description: Complete pathologic response is defined as the absence of detectable malignant cells in the prostatectomy specimen evaluated by standard histologic techniques.
Time Frame: From baseline and time of radical prostatectomy (average of week 9)
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Cohort
Number analyzed (Participants) | 12
Participants | 0

10. Secondary Outcome: Number of Participants With Serologic Response
Description: Best serologic response secondary to immune treatment was reported. Change in Prostate-specific Antigen (PSA) was used to identify serological responses among participants in the lead-in cohort. Complete Serological Response was defined as PSA level less than 0.2 ng/mL measured for 2 consecutive measurements at least 4 weeks apart. Partial Serological Response was defined as decline of PSA at least 50% measured for 2 consecutive measurements at least 4 weeks apart. Serological Progression: Serological progression will only be measured once PSA has risen above 4 ng/mL and this value must be 50% above the PSA level before commencing treatment. Increase in PSA more than 50% of nadir (lowest PSA on treatment). Values must be measured for 2 consecutive measurements at least 2 weeks apart. The date of the first increase will be recorded as progression. Stable disease: not meeting progressive disease (PD) criteria for ≥12 weeks from treatment start.
Time Frame: From baseline throughout study completion, an average of 1.4 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort
Number analyzed (Participants) | 12
Participants
  Complete Serological Response | 1
  Partial Serological Response | 1
  Serological Progressive Disease | 4
  Serological Stable Disease | 6

11. Secondary Outcome: Rate of Biochemical Recurrence After Prostatectomy (Only for Neoadjuvant Cohort)
Description: Biochemical recurrence following radical prostatectomy is defined as at least two prostate-specific antigen (PSA) values that are 0.2 ng/mL or higher.
Time Frame: From time of prostatectomy through study completion, an average of 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort | Neoadjuvant Cohort
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

12. Secondary Outcome: Changes in Magnetic Resonance Imaging (MRI) Secondary to Immune Treatment (Only for Neoadjuvant Cohort)
Description: MRI of the prostate was performed to assess for changes in imaging characteristics of prostate cancer pre and post vaccination. MRI changes secondary to immune treatment is defined as increase or decrease in the size of lesions from baseline (pre-vaccine) measurements. Decrease from baseline to after treatment would represent a positive outcome.
Time Frame: From baseline to closest date to prostatectomy, average on week 9.
Population: 4/12 participants were not analyzed because MRI was not performed due to logistical issues.
Measure: Mean (Full Range); unit: mm
Arm/Group | Neoadjuvant Cohort
Number analyzed (Participants) | 8
mm
  Mean largest lesion measurement at baseline | 16.5 [8 to 24]
  Mean targeted lesion measurement after treatment | 17.3 [9 to 25]

13. Secondary Outcome: Changes in Apparent Diffusion Coefficient (ADC) Mapping, Secondary to Immune Treatment (Only for Neoadjuvant Cohort)
Description: Apparent diffusion coefficient (ADC) mapping in magnetic resonance imaging (MRI) is an indicator of tumor cell density. This outcome aims to capture any changes in ADC within the prostate tissue before and after the treatment administration. ADC changes secondary to immune treatment are defined as increase or decrease in ADC from baseline (pre-treatment) measurements. Low ADC values in tumors reflect areas of cell proliferation, and high ADC values reflects necrotic and acellular areas.
Time Frame: From baseline to closest date to prostatectomy, average on week 9.
Population: 4/12 participants were not analyzed because MRI was not performed due to logistical issues.
Measure: Mean (Standard Deviation); unit: 10^6 mm^2/s
Arm/Group | Neoadjuvant Cohort
Number analyzed (Participants) | 8
10^6 mm^2/s
  Mean ADC value for all measurable lesions at baseline | 1220.6 (218.4)
  Mean ADC value for all measurable lesions after treatment | 1236.1 (244.6)

14. Secondary Outcome: Intraprostatic Treg Cell Infiltration With Cluster of Differentiation 4 (CD4+) and Forkhead Box P3 (FOX-P3) Staining (Only for Neoadjuvant Cohort)
Description: Intraprostatic Treg cell infiltration was measured by computer automated staining analysis pre and post treatment. Quantification will be reported as number of stained cells per mm^2 of tissue.
Time Frame: Baseline and at time of prostatectomy (approximately week 9)
Measure: Median (Inter-Quartile Range); unit: Cell/mm^2 of tissue
Arm/Group | Neoadjuvant Cohort
Number analyzed (Participants) | 12
Cell/mm^2 of tissue
  T regs in the total tissue at baseline | 0.3 [0 to 2.7]
  T regs in the total tissue at prostatectomy | 1.3 [0 to 5.3]
  T regs in the center of the tumor at baseline | 0 [0 to 2.5]
  T regs in the center of the tumor at prostatectomy | 1.5 [0 to 5.25]
  T regs in the invasive margin at baseline | 0 [0 to 0.3]
  T regs in the invasive margin at prostatectomy | 3.5 [0 to 9.75]
  T regs in the normal region at baseline | 0 [0 to 0]
  T regs in the normal region at prostatectomy | 0 [0 to 4.25]

15. Secondary Outcome: Number of Participants With Peripheral Prostate-Specific Antigen (PSA)-Specific T Secondary To Immune Treatment
Description: The number of participants who developed positive PSA-Specific T cell responses secondary to immune treatment will be reported. Peripheral prostatic specific antigen (PSA)-specific T cells at baseline and after therapy were assessed. PSA-specific T cells were those producing cytokine (Interferon gamma (IFNγ), Tumor Necrosis Factor Alpha (TNFα), Interleukin-2 (IL-2) or positive for the degranulation marker cluster of differentiation 107a (CD107a) following in vitro stimulation with PSA-15-mer peptides compared to a negative control peptide pool, measured by intracellular cytokine staining. A positive response will be defined as a >2-fold increase in PSA-specific T cells after therapy compared to baseline.
Time Frame: Weeks 7-10 and 17-22 compared to baseline
Population: 1/12 were not analyzed in the lead-in cohort because there was an insufficient number of viable peripheral blood mononuclear cells (PBMC) to perform the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort | Neoadjuvant Cohort
Number analyzed (Participants) | 11 | 12
Participants
  Participants with PSA-specific T cells at baseline | 2 | 6
  Participants with positive PSA-specific Tcell response 7-10weeks post treatment compared to baseline: number analyzed (Participants) | 11 | 11
  Participants with positive PSA-specific Tcell response 7-10weeks post treatment compared to baseline | 7 | 3
  Participants with positive PSAspecific Tcell response 17-22weeks post treatment compared to baseline: number analyzed (Participants) | 9 | 11
  Participants with positive PSAspecific Tcell response 17-22weeks post treatment compared to baseline | 4 | 5

16. Secondary Outcome: Best Overall Response for Participants With Measurable Disease (Only in the Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort)
Description: The best overall response is the best response recorded from the start of the treatment until disease progression/ recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started) measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: Baseline throughout study completion (average 1.4 years)
Population: 7/12 participants had measurable disease at baseline and were analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort
Number analyzed (Participants) | 7
Participants
  Complete Response | 2
  Partial Response | 0
  Stable Disease | 3
  Progressive Disease | 2

17. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: First study intervention, Study Day 1, to 30 days after participant received last study drug administration. Approximately 1.4 years for the metastatic castration-resistant prostate cancer cohort, and an average of 20 weeks for the neoadjuvant cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort | Neoadjuvant Cohort
Number analyzed (Participants) | 12 | 12
Participants | 12 | 12

ADVERSE EVENTS:
Time Frame: From the first study intervention, Study Day 1, through 30 days after the participant received the last study drug administration. Approximately 1.4 years for the metastatic castration-resistant prostate cancer (mCRPC) cohort, and an average of 20 weeks for the neoadjuvant cohort.
Description: First study intervention, Study Day 1, to 30 days after participant received last study drug administration. Approximately 1.4 years for the metastatic castration-resistant prostate cancer cohort, and an average of 20 weeks for the neoadjuvant cohort.
Arm/Group | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort | Neoadjuvant Cohort
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 6/12 | 3/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort (N=12) | Neoadjuvant Cohort (N=12)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
GGT increased (Investigations) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Immune medicated sicca syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) — Adenocarcinoma of Jejunum
Renal and urinary disorders - Other, Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Lichenoid drug reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Cohort (N=12) | Neoadjuvant Cohort (N=12)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (9) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (6) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 5 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Bloating (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, Amylase increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, Feels hot all the time (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 2 (3) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (4) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
CPK increased (Investigations) | 1 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 1 (1)
Creatinine increased (Investigations) | 3 (4) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Edema limbs (General disorders) | 2 (3) | 1 (2)
Edema trunk (General disorders) | 0 (0) | 1 (2)
Eye disorders - Other, Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (6) | 0 (0)
Fatigue (General disorders) | 7 (14) | 5 (6)
Fever (General disorders) | 3 (3) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (3) | 7 (11)
Gait disturbance (General disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders - Other, Polydipsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, degenerative teeth 22&27 (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Right lower leg edema (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, retching, gagging (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, sweating intermittent (General disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 2 (4)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (3) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (15) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (10) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 12 (75) | 10 (31)
Injury, poisoning and procedural complications - Other, Abrasions left hand (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, Mild head injury (hit his head) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Investigations - Other, Elevated HgbA1c (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 3 (7) | 2 (4)
Lymphocyte count decreased (Investigations) | 2 (10) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, Poor appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (3) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — adenocarcinoma of the jejunum
Nervous system disorders - Other, lightness - positional standing up (Nervous system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (3)
Renal and urinary disorders - Other, UTI (Renal and urinary disorders) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other, Penile lesions (Balanitis) (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Reproductive system and breast disorders - Other, Penile retraction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 2 (7) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash- small circular pinpoint areas of brown and pink flat lesions
Skin and subcutaneous tissue disorders - Other, Right groin incision disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, rash and coating of tongue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, skin rash eyes area and hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, BL ureteral stent exchanges- Annual (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Bilateral stent placements (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) — Bloating, bladder spasm, urinary leakage, bruise R thigh, Scrotal edema, LE edema
Surgical and medical procedures - Other, Esophagogastroduodenoscopy (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Positive Cologuard test (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Small bowel resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Surgical incision (Abdomen) (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Ultrasound guided percutaneous drain for findings of left (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, left percutaneous nephrostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, rt nephro-ureterostomy tube exchange (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 3 (4) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (6) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (2) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Weight loss (Investigations) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT02933255/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT02933255/ICF_001.pdf